CLINICAL TRIAL: NCT04475640
Title: GEMINI - Cancer Genetic Testing in Ethnic Populations
Brief Title: Cancer Genetic Testing in Ethnic Populations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 19-006717; NCI-2020-04427 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-006717 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2020-06-25; First posted 2020-07-17 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Breast Carcinoma; Carcinoma of Unknown Primary; Central Nervous System Carcinoma; Digestive System Carcinoma; Genitourinary System Carcinoma; Head and Neck Carcinoma; Malignant Brain Neoplasm; Malignant Female Reproductive System Neoplasm; Malignant Musculoskeletal Neoplasm; Malignant Solid Neoplasm; Skin Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Neoplasms, Unknown Primary; Brain Neoplasms | interventions — Specimen Handling; Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (biospecimen collection) (Experimental): Patients undergo collection of blood or saliva sample for genetic testing.
  Interventions: Procedure: Biospecimen Collection; Other: Genetic Testing

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood sample
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Genetic Testing — Undergo genetic testing
  Other Names: Genetic Analysis; Genetic Examination; Genetic Test

SUMMARY:
This clinical trial examines the integration of cancer genetic testing in various ethnic populations. Studying individuals and families at risk of cancer may help identify cancer genes and other persons at risk. The information from this study may provide an opportunity for cancer risk stratification and individualized screening in these ethnic populations.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the prevalence of genetic mutations in cancer patients from various ethnic populations seeking care at Mayo Clinic Arizona and Mayo Clinic Florida cancer clinics.

SECONDARY OBJECTIVES:

I. Perform a chart review to assess the impact of genetic testing as part of standard of oncology care:

Ia. Determine prevalence of pathogenic germline mutation detected by multi-gene panel testing.

Ib. Determine differences in germline mutation detection in these patients as compared to traditional guideline (National Comprehensive Cancer Network [NCCN]) based approach for genetic evaluation.

OUTLINE:

Patients undergo collection of blood or saliva sample for genetic testing.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age
* Individuals diagnosed with any solid tumor cancer including, but not limited to, gastrointestinal, breast, gynecological, genitourinary, skin, central nervous system (CNS)/brain, head/neck, musculoskeletal or cancer of unknown primary; and presenting to Mayo Clinic (MC Arizona or MC Florida) for clinical management/treatment; and patients receive genetic testing as described above
* Self-identified as being from various ethnic populations including Hispanic/Latino, Native American/Alaskan, African American (including of African descent), Asian and other European populations
* Blood collection is feasible (health, access and/or tolerability) for requested blood sample(s)
* Individuals have agreed to participate and signed the study informed consent form

Exclusion Criteria:

* Patients who have had prior germline genetic testing involving a 40+ gene panel within the last 24 months at Mayo Clinic and available for review by the research coordinator at time of consent
* Past or current history of hematological cancer (including leukemias, multiple myeloma)
* All bone marrow transplants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2020-01-13 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Prevalence of pathogenic germline mutations in enrolled patients within each cancer site | Study completion (2 years)
  Will identify the prevalence of pathogenic germline mutations in enrolled patients within each cancer site, age (< 60 years old versus (vs.) >= 60 years old), and stage (early vs. advanced) via descriptive statistics.
Prevalence of positive pathogenic germline mutations | Study completion (2 years)
  Will determine whether the prevalence of positive pathogenic germline mutations differs between cancer sites, age of diagnosis, and stage of diagnosis using logistic regression analysis across all cancer site groups and pairwise post-hoc analyses using Tukey's correction for multiple comparisons across pairs of cancer sites and chi-square tests of differences between age and stage groups.
Rate of mutation detection via genetic testing to clinical practice guidelines of traditional family history criteria | Study completion (2 years)
  Will compare the rate of mutation detection via genetic testing to clinical practice guidelines of traditional family history criteria within cancer site, age, and stage using logistic regression and pairwise post-hoc analyses as needed.
Impact of germline genetic testing on both therapeutic management and targeted cancer prevention | Study completion (2 years)
  Will assess the impact of germline genetic testing on both therapeutic management and targeted cancer prevention in family members using logistic regression and pairwise post-hoc analyses as needed.

CONTACTS AND LOCATIONS:
Overall Officials: Jewel Samadder, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials